CLINICAL TRIAL: NCT02983435
Title: Comparison Between Two Osteopathic Techniques for Chronic Low Back Pain Treatment: a Randomized Crossover Trial.
Brief Title: Osteopathic Treatment for Chronic Low Back Pain
Acronym: OTCLBP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Norte do Paraná (Other)
Responsible Party: Principal Investigator, Rubens Alexandre da Silva Jr, Professor, Universidade Norte do Paraná
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: rubens@unopar.br
Record Dates: First submitted 2016-11-25; First posted 2016-12-06 (Estimated); Last update posted 2018-09-07 (Actual); Status verified 2018-09

CONDITIONS: Low Back Pain; Osteopathic Manipulative Treatment
Keywords: Osteopathic Treatment; Postural control; Neuromuscular activation; Physiotherapy
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- G1 - Thrust manipulation (Experimental): G1 - Thrust manipulation is an osteopathic technique. The Group 1 (G1) will receive the Thrust technique applied at the level of dysfunction. Subject in lateral decubitus, with one lower limb extended and the other in flexion, to the level of the targeted vertebra; upper trunk rotated back until the same vertebra; at the end of the range of movement will be applied the high speed and low amplitude impulse (Thrust).
  Interventions: Other: G1 - Thrust manipulation
- G2 - Muscle Energy (Active Comparator): G2 - Muscle Energy is a manual therapy technique based in muscular contraction and stretching. The Group 2 (G2) will receive the Muscle Energy technique applied at the level of dysfunction. Subject in lateral decubitus, with the upper and lower trunk flexed until the target vertebra, and upper trunk rotated back to the level of the same vertebra; lumbar in lateral flexion (using the subject's feet) until the target vertebra. Following the command the subject will perform an isometric contraction of 3-5 seconds against the therapist's hand (pushing the hand towards the floor), repeated 3 times.
  Interventions: Other: G2 - Muscle Energy

INTERVENTIONS:
Other: G1 - Thrust manipulation — Osteopathic manipulation with Thrust technique. The Group 1 (G1) will receive the Thrust technique applied at the level of dysfunction. Subject in lateral decubitus, with one lower limb extended and the other in flexion, to the level of the targeted vertebra; upper trunk rotated back until the same vertebra; at the end of the range of movement will be applied the high speed and low amplitude impulse (Thrust).
  Arms: G1 - Thrust manipulation
Other: G2 - Muscle Energy — Osteopathic manipulation with Muscle Energy technique. The Group 2 (G2) will receive the Muscle Energy technique applied at the level of dysfunction. Subject in lateral decubitus, with the upper and lower trunk flexed until the target vertebra, and upper trunk rotated back to the level of the same vertebra; lumbar in lateral flexion (using the subject's feet) until the target vertebra. Following the command the subject will perform an isometric contraction of 3-5 seconds against the therapist's hand (pushing the hand towards the floor), repeated 3 times.
  Arms: G2 - Muscle Energy

SUMMARY:
The relevance of this study is to determine the efficacy of two osteopathic techniques - Thrust Technique and Muscle Energy Technique (MET) - in improving of neuromuscular component of the trunk and clinical symptoms in adult workers with Chronic Low Back Pain (CLBP). Few studies have investigated and compared the physiological responses of these techniques quantitatively, and no published study has compared their effects in low back pain subjects in terms of symptoms, postural balance and muscle activation. The main outcomes will be computed by electromyography measurement so that to assess the trunk neuromuscular activation pattern as well as by force platform parameters for determining of postural control. Clinical symptoms such as pain intensity, perception of disability and fear and avoidance will also be computed.

This is the first study to compare these two osteopathic techniques using the main biological outcomes related to trunk neuromuscular function.

DETAILED DESCRIPTION:
The purpose of this study is to assess the efficacy of two osteopathic techniques (Thrust and MET) on CLBP adult workers treatment.

A total of 15 male participants with chronic low back pain, volunteers, active workers aged from 35 to 55 years (in aging process) will be recruited by convenience from the community local. All participants will sign an informed consent form approved by the North of Parana University Ethics Committee for Research on Human Subjects. The intervention will follow the CONSORT recommendations for randomized controlled trials. All baseline testing and evaluation will be performed by a blinded evaluator to the study intervention. The sample will be randomized in two groups from crossover design: Group #1), which will receive the Thrust technique applied at the level of dysfunction; and Group #2, which will receive the Muscle Energy Technique, also applied at the level of dysfunction. The allocation will be printed in cards by sequentially numbered in opaque envelopes.

The treatment (intervention) will occur in 2 phases of 3 weeks each one. The participants will receive only one of techniques in each phase, and after one rest week (washout) they will receive the other technique (crossover), totaling 7 weeks. In this study, both techniques will be applied at the lumbar vertebral level that present the dysfunction which will be diagnosed in the specific evaluation, performed by two specialized physiotherapists in osteopathy. Before and after the manipulation (with Thrust or MET) all participants will be evaluated in 2 tasks - bipedal without load and bipedal with load (10% of body mass) - on the force platform. Parallel to the tasks, the recording of the measurements of EMG surface will be computed to determine the pattern of the trunk neuromuscular activation in amplitude of the RMS signal as well as muscle fatigue through the median frequency parameters.

Before performing the tasks on the force platform, a maximum voluntary isometric contraction will be performed for the back (paravertebral) and abdominal (rectus) muscles in order to normalize the signal EMG for determining of the level muscular activity during each task (with or without load). After the intervention, the immediate and final revaluations will include all the used measures in the initial evaluation, such as muscle activation of trunk (EMG), balance (force platform), and clinical symptoms of pain (Visual Analogue Scale and McGill Short Questionnaire), psychosomatic factors (Fear and Avoidance Believe Questionnaire) and disability (Roland Morris Questionnaire).

For the analysis a two-way ANOVA will be used for each dependent variable to compare the two groups (G1 versus G2) in both situations (pre and post-immediate, and after 15 days) in the clinical measurements, postural balance and EMG. The size effect also will be computed to determine the rate of the changes observed.

ELIGIBILITY:
Inclusion Criteria:

* Chronic low back pain at least for three months.
* Low back pain of unknown mechanical origin without irradiation to the lower limbs.
* Workers with chronic low back pain at least three months.
* Do not be participating in rehabilitation programs.
* Do not have practiced regular physical activity in the past 3 months.

Exclusion Criteria:

* Manual therapy treatment in the past 90 days.
* Discal herniation diagnosis.
* Lumbar radiculopathy and / or nerve root compression.
* Lumbar stenosis.
* Lumbar surgery.
* Nerve root entrapment.
* Neurological and endocrine.
* Osteoporosis.
* Rheumatoid arthritis.
* Spinal osteomyelitis.
* Spondylolysis.
* Spondylolisthesis.
* Tumors.
* Vertebral fracture.
* No current sports or treatment in Physiotherapy, Pilates Method or Manual Therapy.

Ages: 35 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2016-12; Primary Completion 2017-03 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Electromyography measurement - Root Mean Square (RMS) | Change from baseline muscular activation at 3 weeks, in both phases
  EMG estimates, Root Mean Square: RMS (in microvolts unit: uV) will be computed to evaluate the back and abdominal activation during the functional task.

SECONDARY OUTCOMES:
Electromyography measurement - Median Frequency (MF) | Change from baseline muscular activation at 3 weeks, in both phases
  EMG estimates, Median Frequency: MF (in Hertz: Hz) will be computed to evaluate the back and abdominal activation during the functional task.
Force platform measurement | Change from baseline muscular activation at 3 weeks, in both phases
  Force platform measurement during balance performance using centre of pressure measures to assess balance performance.

OTHER OUTCOMES:
Visual Analogic Scale | Change from baseline muscular activation at 3 weeks, in both phases
  Pain intensity measurement using Visual Analogue Scale (score of 0 to 10 intensity; being 10 of poor score for VAS).
Short Version of Pain Questionnaire McGill | Change from baseline muscular activation at 3 weeks, in both phases
  Pain measurement using Short Version of Pain Questionnaire McGill (score 0 to 78; while higher score is determined by poor condition related to pain).
Disability questionnaire | Change from baseline muscular activation at 3 weeks, in both phases
  Disability measurement using Roland Morris questionnaire.
Fear-avoidance questionnaire | Change from baseline muscular activation at 3 weeks, in both phases
  Fear-avoidance model measurement using Waddell questionnaire related to work and physical activity.

CONTACTS AND LOCATIONS:
Overall Officials: Rubens da Silva, PhD, Study Director — Laboratory of Functional Assessment and Human Motor Performance (LAFUP)
Locations (1):
- Laboratory of Functional Assessment and Human Motor Performance (LAFUP), Londrina, Paraná, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Licciardone JC, Minotti DE, Gatchel RJ, Kearns CM, Singh KP. Osteopathic manual treatment and ultrasound therapy for chronic low back pain: a randomized controlled trial. Ann Fam Med. 2013 Mar-Apr;11(2):122-9. doi: 10.1370/afm.1468. PMID 23508598
- [Background] Haas M, Vavrek D, Peterson D, Polissar N, Neradilek MB. Dose-response and efficacy of spinal manipulation for care of chronic low back pain: a randomized controlled trial. Spine J. 2014 Jul 1;14(7):1106-16. doi: 10.1016/j.spinee.2013.07.468. Epub 2013 Oct 16. PMID 24139233
- [Background] Wilder DG, Vining RD, Pohlman KA, Meeker WC, Xia T, Devocht JW, Gudavalli RM, Long CR, Owens EF, Goertz CM. Effect of spinal manipulation on sensorimotor functions in back pain patients: study protocol for a randomised controlled trial. Trials. 2011 Jun 28;12:161. doi: 10.1186/1745-6215-12-161. PMID 21708042
- [Background] Cleland JA, Fritz JM, Childs JD, Kulig K. Comparison of the effectiveness of three manual physical therapy techniques in a subgroup of patients with low back pain who satisfy a clinical prediction rule: study protocol of a randomized clinical trial [NCT00257998]. BMC Musculoskelet Disord. 2006 Feb 10;7:11. doi: 10.1186/1471-2474-7-11. PMID 16472379
- [Background] da Silva RA Jr, Arsenault AB, Gravel D, Lariviere C, de Oliveira E Jr. Back muscle strength and fatigue in healthy and chronic low back pain subjects: a comparative study of 3 assessment protocols. Arch Phys Med Rehabil. 2005 Apr;86(4):722-9. doi: 10.1016/j.apmr.2004.08.007. PMID 15827924
- [Background] Lariviere C, Gagnon D, Loisel P. The comparison of trunk muscles EMG activation between subjects with and without chronic low back pain during flexion-extension and lateral bending tasks. J Electromyogr Kinesiol. 2000 Apr;10(2):79-91. doi: 10.1016/s1050-6411(99)00027-9. PMID 10699556